CLINICAL TRIAL: NCT06087029
Title: IMPRoving Outcomes in Vascular DisEase- Aortic Dissection
Brief Title: IMPRoving Outcomes in Vascular DisEase - Aortic Dissection
Acronym: IMPROVE-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); State University of New York - Downstate Medical Center (Other); Oregon Health and Science University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00113329; 4UH3HL165017-02 (NIH); 5U24HL165029-02 (NIH)
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Type B Aortic Dissection
Keywords: TEVAR
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront TEVAR plus Medical Therapy (Experimental): Participants randomized to upfront TEVAR will receive a commercially available device customized to their individual anatomical requirements. Stent-graft implantation will be performed either in the operating room with appropriate digital imaging equipment to allow fluoroscopic and trans-esophageal echo (TEE) guidance or the catheterization laboratory, angiographic suite (with digital angiographic equipment).
  Interventions: Procedure: TEVAR; Other: Guideline directed medical therapy and surveillance of dissection
- Medical Therapy with surveillance for deterioration (Active Comparator): Participants randomized to upfront Medical Therapy with Surveillance for Deterioration will be treated per routine clinical care with suggested antihypertensive therapy and cardiovascular risk factor reduction as per appropriate cardiovascular guidelines.
  Interventions: Other: Guideline directed medical therapy and surveillance of dissection

INTERVENTIONS:
Procedure: TEVAR — Thoracic endovascular aortic repair
  Arms: Upfront TEVAR plus Medical Therapy
Other: Guideline directed medical therapy and surveillance of dissection — Routine clinical care with suggested antihypertensive therapy and cardiovascular risk factor reduction as per appropriate cardiovascular guidelines.

SUMMARY:
The goal of this clinical trial is to determine whether an upfront invasive strategy of TEVAR plus medical therapy reduces the occurrence of a composite endpoint of all-cause death or major aortic complications compared to an upfront conservative strategy of medical therapy with surveillance for deterioration in patients with uncomplicated type B aortic dissection.

DETAILED DESCRIPTION:
The study will be a prospective, pragmatic, randomized clinical trial of the comparative effectiveness of an initial strategy for the treatment of uncomplicated type B aortic dissection (uTBAD). Patients with uTBAD and no prior history of aortic intervention will be randomized within 48 hours to 6 weeks after index admission to one of the two initial strategies. Follow-up will be ascertained via a centralized call center and ascertainment of medical records, as well as remote blood pressure monitoring. Recommendations regarding medical therapy will be made to enrolling centers and feedback on the quality of medical care given, however, all subsequent care, with the exception of aortic interventions, will be at the discretion of the responsible clinical care team. Aortic interventions will allowable only as per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years
2. Patients with a Stanford type B aortic dissection not involving the aorta at or proximal to the innominate artery, without rupture and/or malperfusion syndrome (renal, mesenteric, or extremity) who are within 48 hours to 6 weeks after start of index admission for their type B dissection

4. Ability to provide written informed consent 5. Investigator believes anatomy is suitable for TEVAR

Exclusion Criteria:

1. Ongoing systemic infection
2. Pregnant or planning to become pregnant in the next 3 months
3. Life expectancy related to non-aortic conditions < 2 years
4. Unwilling or unable to comply with all study procedures
5. Known patient history of genetic aortopathy
6. Penetrating Aortic Ulcer without concomitant uTBAD
7. Intramural hematoma without concomitant uTBAD
8. Iatrogenic (traumatic) aortic dissection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause death or major aortic complications (MAC) | Last follow-up timepoint. Differential follow-up with median of about 4 years
  The primary endpoint is a composite of all-cause death or major aortic complications (MAC). MACs are defined as:
  * Aortic rupture
  * Malperfusion syndrome
  * New aortic tear requiring intervention,
  * Retrograde aortic dissection,
  * Dependence on outpatient dialysis (chronic)
  * Major amputation (above ankle)
  * Tracheostomy
  * fistula formation (e.g., aorto-esophageal, aorto-tracheal)
  * Spinal Cord Ischemia with paralysis or paresis
  * Stroke
  * AD-related intervention in either group defined as:
    * Open TAA/TAAA Repair
    * Fenestrated and/or Branched Endovascular Repair of TAAA
    * Repeat TEVAR

SECONDARY OUTCOMES:
Quality of Life, as measured by the Abdominal Aortic Aneurysm Quality of Life questionnaire (AAAQol) | Last follow-up timepoint. Differential follow-up with median of about 4 years
  An adapted version of the AAAQol survey and the PROMIS-16 will be used to assess general and aortic specific quality of life. The AAAQol questionnaire was specifically developed and validated on patients with abdominal aortic aneurysms and measures both the physical and emotional impact of either 1) having an abdominal aortic aneurysm or 2) having surgical or endovascular therapy for an abdominal aortic aneurysm. This metric has been shown to be valid and responsive in abdominal aortic aneurysm. While it has not been tested in aortic dissection, its questions assess the same domains shown to be significantly impacted in patients with aortic dissection.
Cumulative incidence of cardiovascular (CV) hospitalizations | Last follow-up timepoint. Differential follow-up with median of about 4 years
  CV hospitalization will be defined as hospitalization >/= 24 hours for any cardiovascular cause.
Mean number of cardiovascular (CV) hospitalizations | Last follow-up timepoint. Differential follow-up with median of about 4 years
  CV hospitalization will be defined as hospitalization >/= 24 hours for any cardiovascular cause.
Incidence of cardiovascular death | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Death from any cardiovascular cause.
Incidence of all-cause death | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Death from any case
Cumulative incidence of major aortic complications (MAC) | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Composite endpoint. MACs are defined as: • Aortic rupture • Malperfusion syndrome • New aortic tear requiring intervention, • Retrograde aortic dissection, • Dependence on outpatient dialysis (chronic) • Major amputation (above ankle) • Tracheostomy • fistula formation (e.g., aorto-esophageal, aorto-tracheal) • Spinal Cord Ischemia with paralysis or paresis • Stroke • AD-related intervention in either group defined as: - Open TAA/TAAA Repair - Fenestrated and/or Branched Endovascular Repair of TAAA - Repeat TEVAR
Incidence of stroke | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Defined as a focal neurological deficit that could be attributed to a vascular territory and lasted >24 hours or was associated with a new lesion on computed tomography scan or magnetic resonance imaging.
Incidence of paraplegia or paraparesis | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Defined as including: 1) flaccid paraplegia (no lower extremity movement), or lower extremity movement without gravity, or lower extremity movement with gravity, or standing with assistance or walking with assistance.
Incidence of vascular access injury requiring surgical repair | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Defined as any open surgical procedure to treat a vascular injury at the site of vascular access for a previous endovascular procedure.
Incidence of aortobronchial / aortoesophageal fistula | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Defined as fistulous connection between the aorta and bronchus as confirmed by chest imaging or direct visualization (surgical or bronchoscopic). Aortoesophageal fistula is defined as a fistulous connection between the aorta and the esophagus as confirmed by chest imaging or direct visualization (surgical or endoscopically).
Incidence of retrograde type A dissection | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Defined as any new ascending arch, or descending dissection contiguous with and proximal to the original presenting anatomy as confirmed by imaging.
Incidence of aortic-related death | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Aortic-related death will be defined as death within 30 days of 1) diagnosis of aortic dissection 2) any aortic intervention or 3) ruptured aortic aneurysm.
Number of days alive and out of the hospital | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Defined as the number of days alive minus the number of days in the hospital over 4 years (primary analysis).
Incidence of secondary percutaneous interventions after TEVAR | Last follow-up timepoint. Differential follow-up with median of about 4 years
  Any secondary percutaneous intervention after TEVAR

CONTACTS AND LOCATIONS:
Overall Officials: Manesh R Patel, M.D., Principal Investigator — Duke University; Firas F Mussa, M.D., Principal Investigator — The University of Texas at Houston; Panos Kougias, M.D., Principal Investigator — The State University of New York at Downstate; Sreekanth Vemulapalli, M.D., Principal Investigator — Duke University; Sean O'Brien, Ph.D., Principal Investigator — Duke University
Locations (60):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Honorhealth, Phoenix, Arizona
  - Memorial Care Long Beach Medical Center, Long Beach, California
  - Keck Medical Center of USC, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of California, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Florida Health, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - MaineHealth, Scarborough, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial, Worcester, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health and Hospitals and Corewell, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Rutgers UH Vascular Center, Newark, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - St. Francis Hospital and Heart Center, Roslyn, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Sanger Heart & Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Harrington Heart and Vascular Institute, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Dell Medical School- Ascension, Austin, Texas
  - Baylor Scott & White Research Institution, Dallas, Texas
  - UT Southwestern- Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Houston, Houston, Texas
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The Statistical and data analytic center (SDCC) will submit to the NHLBI data repository de-identified Limited Access Datasets (LADs) and associated documentation, for use by other investigators. The LADs and documentation will be submitted within 2 years after publication of the primary results manuscript. Documentation will include copies of the case report forms; a list of derived variables and the formulas used to create them; and a codebook providing for each variable the variable name, coding conventions, and distribution of values. It will also include a list of data modifications made when creating the LAD, and a copy of the informed consent template, so that future use of the data will be consistent with the consent provided by the study subjects.The goal is to make data available to other investigators while protecting the rights and privacy of the subjects who participated in the studies. The SDCC will anonymize the datasets.
Supporting Information: ICF
Time Frame: 2 years
Access Criteria: The methods for restricting access will also need to be determined, either with password access and/or with executed Data Agreements. Related to the restricted use of data is the need to specify appropriately in informed consent forms that the study participant's de-identified data may be made available to other researchers.